CLINICAL TRIAL: NCT01452230
Title: Effectiveness and Efficacity of Presurgery Supervised Physical Activity Training on Health of Obese Individuals Waiting for Bariatric Surgery
Brief Title: Prebariatric Surgery Physical Activity Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Marie-France Langlois, Principal investigator, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 11-112
Record Dates: First submitted 2011-10-07; First posted 2011-10-14 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Obesity
Keywords: Bariatric Surgery Candidate; Severely obese; Bariatric surgery; Physical activity; Physical fitness; Comorbidities; Quality of life; Surgical complications
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supervised physical activity (Experimental)
  Interventions: Behavioral: Supervised physical activity
- Usual care (No Intervention)

INTERVENTIONS:
Behavioral: Supervised physical activity — Supervised physical activity
  Arms: Supervised physical activity

SUMMARY:
Introduction: According to studies, a low physical capacity before surgery is linked with smaller weigh loss after surgery and increases risks of peri-surgical complications. Practice of regular physical activity in obese individuals improves their physical capacity. No specific recommendation on physical activity prescription is currently available for this reduced fitness population. This project aims to evaluate if a Pre-Surgical Physical Activity Training (PreSPAT) improves physical capacity, surgery effectiveness and decreases peri-surgical complications in morbidly obese individuals.

Methods: This pilot project will be divided in 2 phases:

Phase 1: Ten candidates for bariatric surgery will be included in this phase. In a pre-training focus group, subjects will be interviewed about their expectations and their availability for a PreSPAT. These results combined with those of the literature will be used to design the PreSPAT. To measure its effectiveness, anthropometric parameters, body composition, physical capacity, motivational stage, perceived benefits and barriers facing physical activity and quality of life will be evaluated before and after the PreSPAT. Subjects satisfaction with the physical activity intervention will be measured with a questionnaire at 6 weeks and at the end of the PreSPAT.

Phase 2: 50 candidates for bariatric surgery will be randomized in 2 groups:

Control group: receiving usual care from the integrated medical and surgical treatment obesity clinic of the Centre Hospitalier Universitaire de Sherbrooke, which includes individual counselling by an exercise physiologist every 6 weeks.

Intervention group: will attend for three months before surgery sessions of supervised physical activity as developed during phase 1 in addition to usual care of the integrated medical and surgical treatment obesity clinic.

Physical capacity, anthropometry, body composition, readiness to change, comorbidities, perceived benefits and barriers of physical activity, usual practice of physical activity, quality of life and patient satisfaction with physical activity intervention will be evaluated in the two groups before and after intervention and every 3 months after the surgery during one year. Each occurrence of peri-surgery complications, and the duration of surgery and hospitalization will be recorded.

Impacts: Feasibility and effectiveness of supervised physical activity training will be assessed before the beginning of the randomized controlled study. Phase 2 of the project may generate information that will improve the management of obese candidates for bariatric surgery in order to ensure optimal results for their health. This project will also allow a better understanding of criteria leading to successful surgery and the effects of exercise training in morbidly obese individuals.

DETAILED DESCRIPTION:
Introduction: Bariatric surgery appears to be the most effective solution to improve health in morbidly obese individuals. However, this intervention is associated with risks than could be lower with pre-surgery intervention. According to studies, a low physical capacity before surgery is linked with smaller weigh loss after surgery and increases risks of peri-surgical complications. Practice of regular physical activity in obese individuals improves their physical capacity. No specific recommendation on physical activity prescription is currently available for this reduced fitness population. This project aims to evaluate if a Pre-Surgical Physical Activity Training (PreSPAT) improves physical capacity, surgery effectiveness and decreases peri-surgical complications in morbidly obese individuals. Hypotheses: In bariatric surgery patients, the PreSPAT should improve:

* subjects'health (physical capacity, weight, comorbidities, quality of life)
* subjects' motivation to do regular physical activity, their perceived benefits and barriers to do physical activity including pain, discomfort and dyspnea and their satisfaction with their physical activity management
* the duration of surgery and complications
* the postoperative management (duration, complications, re-operation, re-hospitalization). These two last items will probably require a larger population in a future project to complete data if they are conclusive.

Materials and methods: This pilot project will be divided in 2 phases:

Phase 1: Ten candidates for bariatric surgery will be included in this phase. In a pre-training focus group, subjects will be interviewed about their expectations and their availability for a PreSPAT. These results combined with those of the literature will be used to design the PreSPAT. To measure its effectiveness, anthropometric parameters, body composition, physical capacity, motivational stage, perceived benefits and barriers facing physical activity and quality of life will be evaluated before and after the PreSPAT. Subjects satisfaction with the physical activity intervention will be measured with a questionnaire at 6 weeks and at the end of the PreSPAT.

Phase 2: 50 candidates for bariatric surgery will be randomized in 2 groups:

Control group: receiving usual care from the integrated medical and surgical treatment obesity clinic of the Centre Hospitalier Universitaire de Sherbrooke, which includes individual counselling by an exercise physiologist every 6 weeks.

Intervention group: will attend for three months before surgery sessions of supervised physical activity as developed during phase 1 in addition to usual care of the integrated medical and surgical treatment obesity clinic.

Physical capacity, anthropometry, body composition, readiness to change, comorbidities, perceived benefits and barriers of physical activity, usual practice of physical activity, quality of life and patient satisfaction with physical activity intervention will be evaluated in the two groups before and after intervention and every 3 months after the surgery during one year. Each occurrence of peri-surgery complications, and the duration of surgery and hospitalization will be recorded.

Impacts: Feasibility and effectiveness of supervised physical activity training will be assessed before the beginning of the randomized controlled study. Phase 2 of the project may generate information that will improve the management of obese candidates for bariatric surgery in order to ensure optimal results for their health. This project will also allow a better understanding of criteria leading to successful surgery and the effects of exercise training in morbidly obese individuals.

ELIGIBILITY:
Inclusion Criteria:

* bariatric surgery candidate : morbid obesity (BMI>40)or severe obesity (BMI>35 with complications)
* > 18 years old
* follow usual care in the "Clinique médico-chirurgicale du traitement de l'obésité du Centre Hospitalier Universitaire de Sherbrooke (CHUS)" and ready to do presurgery evaluation(approximately 3 month before surgery)
* no regular supervised physical activity
* be willing to do on site supervised physical activity training
* have read and given consent

Exclusion Criteria:

* impossibility to come regularly to the CHUS to participate in physical activity training
* medical contraindication for physical activity
* major functional limitations: failure to realize the 6 minutes walking test
* intellectual disability and / or neuropsychological disease
* not being able to speak or understand french
* being in Prochaska pre contemplation stage for regular physical activity practice

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-10; Primary Completion 2015-06 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in physical fitness 2 weeks before surgery | 2 weeks before surgery

SECONDARY OUTCOMES:
Change from baseline in quality of life 2 weeks before surgery and every 3 months post surgery | 2 weeks before surgery and every 3 months post surgery for 1 year
Number of participants with peri-operative complications | every 3 months post surgery for 1 year
Change from baseline in comorbidities 2 weeks before surgery | 2 weeks before surgery
Number of patients who did lifestyle modification | 2 weeks before surgery and every 3 months post surgery for 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Marie-France Langlois, MD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec, Canada

REFERENCES:
- [Derived] Baillot A, Vallee CA, Mampuya WM, Dionne IJ, Comeau E, Meziat-Burdin A, Langlois MF. Effects of a Pre-surgery Supervised Exercise Training 1 Year After Bariatric Surgery: a Randomized Controlled Study. Obes Surg. 2018 Apr;28(4):955-962. doi: 10.1007/s11695-017-2943-8. PMID 28963710
- [Derived] Baillot A, Mampuya WM, Dionne IJ, Comeau E, Meziat-Burdin A, Langlois MF. Impacts of Supervised Exercise Training in Addition to Interdisciplinary Lifestyle Management in Subjects Awaiting Bariatric Surgery: a Randomized Controlled Study. Obes Surg. 2016 Nov;26(11):2602-2610. doi: 10.1007/s11695-016-2153-9. PMID 27038045